CLINICAL TRIAL: NCT02658188
Title: Long-term Study - Long-term Efficacy and Safety of Gabapentin Enacarbil in Japanese Restless Legs Syndrome Patients
Brief Title: Long-term Efficacy and Safety of Gabapentin Enacarbil in Japanese Restless Legs Syndrome Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8825-CL-0005
Record Dates: First submitted 2016-01-13; First posted 2016-01-18 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-02

CONDITIONS: Restless Legs Syndrome
Keywords: Restless legs syndrome patients; ASP8825; XP13512
MeSH Terms: conditions — Restless Legs Syndrome | interventions — 1-(((alpha-isobutanoyloxyethoxy)carbonyl)aminomethyl)-1-cyclohexaneacetic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ASP8825 group (Experimental)
  Interventions: Drug: ASP8825

INTERVENTIONS:
Drug: ASP8825 — Oral
  Other Names: gabapentin enacarbil

SUMMARY:
The objective of this study is to evaluate the efficacy and safety of ASP8825 (gabapentin enacarbil) for long-term treatment of restless legs syndrome patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients who diagnosed with RLS according to the diagnostic criteria established by the International RLS Study Group
* International Restless Legs Syndrome Scale (IRLS) score ≥15 presence of RLS symptoms on ≥15 days per month and ≥4 days per week preceding inclusion in this study

Exclusion Criteria:

* Patients using dopamine agonists or gabapentin within 1 week before or any anti-RLS treatment within 2 weeks before the start of the pretreatment observation period
* Patients with an estimated creatinine clearance <60 mL/min determined using the Cockcroft-Gault formula
* Pregnant or lactating women
* Individuals with serum ferritin <20 ng/mL were also excluded from the trial
* Individuals with movement disorders and/or abnormal neurological findings

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2007-12; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in IRLS score | Baseline to Week 52
  IRLS: International Restless Legs Syndrome Scale
Safety assessed by Vital signs | Up to Week 52
  Blood pressure and pulse rate
Safety assessed by Adverse Events | Up to Week 52
Safety assessed by Laboratory tests | Up to Week 52
  Hematology, blood biochemistry, thyroid function test and urinalysis
Safety assessed by 12-lead-electrocardiogram | Up to Week 52

SECONDARY OUTCOMES:
Proportion of responders on ICGl of improvement | Up to Week 52
  ICGI: Investigator-rated Clinical Global Impression of improvement
Proportion of responders on PCGI of improvement | Up to Week 52
  PCGI: Patient-rated Clinical Global Impression
Change from baseline in PSQI | Baseline to Week 52
  PSQI: Pittsburgh Sleep Quality Index
Change from baseline in SF-36v2 | Baseline to Week 52
  SF-36v2: Medical Outcomes Study 36-Item Short-Form Health Survey version 2
Change from baseline in RLS-QOL | Baseline to Week 52
  RLS-QOL: Restless Legs Syndrome Quality of Life Questionnaire
Change from baseline in MOS sleep scale | Baseline to Week 52
  MOS: Medical outcomes study
Plasma concentration of gabapentin | Week 12, 28 and 52

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (10):
- Japan (10):
  - Chiba
  - Fukuoka
  - Hokkaido
  - Hyōgo
  - Kanagawa
  - Kyoto
  - Miyagi
  - Osaka
  - Saitama
  - Tokyo

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Link to results on Astellas Clinical Study Results Web site — https://www.astellasclinicalstudyresults.com/hcp/study.aspx?ID=8825-CL-0005